CLINICAL TRIAL: NCT07135414
Title: Accelerated Repetitive Transcranial Magnetic Stimulation in Hospitalized Patients With Obsessive-Compulsive Disorder: a Feasibility and Mechanistic RCT
Brief Title: Accelerated rTMS in Hospitalized Patients With OCD: a Feasibility and Mechanistic Study
Acronym: arTMS-OCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Principal Investigator, Dienstpsychiatrie, Prof. Dr. Chris Baeken, University Hospital, Ghent
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ONZ-2022-0372 AM02 dd 07-Mar-2
Record Dates: First submitted 2025-07-24; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Obsessive - Compulsive Disorder
Keywords: OCD; TMS; deep TMS; iTBS; Obsessive Compulsive Disorder; Transcranial Magnetic Stimulation; OCD-TMS; Hospitalized; Hospitalised; dTMS
MeSH Terms: conditions — Compulsive Personality Disorder; Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial (RCT)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Family and relatives of the patient also remain unaware of the treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- dTMS + ERP (Experimental): 20 hospitalized patients who will receive deep TMS treatment with H7 coil next to psychofarmacological treatment and exposure responseprevention for OCD.
  Interventions: Procedure: dTMS; Behavioral: ERP
- iTBS + ERP (Experimental): 20 hospitalized patients who will receive a specific form of repetitive transcranial magnetic stimulation: intermittent thetaburst stimulation (iTBS) with F8 coil; next to psychofarmacological treatment and exposure responseprevention for OCD.
  Interventions: Procedure: iTBS; Behavioral: ERP
- Control (ERP) (Active Comparator): 20 hospitalized patiënts who will receive psychofarmacological treatment and exposure responseprevention for OCD. No TMS.
  Interventions: Behavioral: ERP

INTERVENTIONS:
Procedure: iTBS — Intermittent theta burst stimulation (iTBS) targeting the left Dorsolateral Prefrontal Cortex (LDLPFC) will be delivered using a figure-of-eight coil at 50 Hz (3 pulses per burst, 5 Hz burst frequency), with 10 bursts over 2 seconds, followed by an 8-second pause, resulting in a 10-second cycle duration, repeated 60 times for a total of 1800 pulses.
  Arms: iTBS + ERP
Procedure: dTMS — Deep TMS (dTMS) targeting the medial prefrontal cortex (MPFC) will be delivered using an H7 coil at 20 Hz for 2 seconds per cycle, followed by a 20-second pause, resulting in a 22-second cycle duration, repeated 50 times for a total of 2000 pulses.
  Arms: dTMS + ERP
Behavioral: ERP — Patients are admitted to a residential program that includes nonverbal therapies, cognitive behavioural therapy, and from week 3 onward, weekly Exposure Relapse Prevention (ERP) sessions (3 hours/week for 8 weeks; total admission = 10 weeks). ERP includes an inventory of OCD symptoms, psychoeducation on the difference between obsessions and compulsions using an OCD model, and the creation of a stepwise fear hierarchy with exposure and response prevention exercises. Patients practice both during and outside sessions, including at home on weekends. Family involvement is integrated: relatives are invited every three weeks to receive psychoeducation on OCD and ERP, are informed about accommodation behaviors, and may attend a session.

SUMMARY:
This study investigates a new treatment approach for Obsessive-Compulsive Disorder (OCD), a condition characterized by unwanted repetitive thoughts and behaviors. The goal is to determine whether combining specialized inpatient care with repetitive Transcranial Magnetic Stimulation (rTMS) is feasible, well-tolerated, and effective. rTMS is a non-invasive procedure that uses magnetic pulses to stimulate specific areas of the brain. In this study, two types of rTMS will be tested: deep TMS (dTMS) and intermittent theta burst stimulation (iTBS). Both treatments will be administered using an accelerated protocol, involving multiple sessions per day over a two-week period.

Patients will be randomly assigned to one of three groups: two groups will receive either dTMS or iTBS combined with Exposure and Response Prevention (ERP), a recognized psychotherapy for OCD; the third group will receive only ERP without rTMS.

Participant Requirements next to treatment:

Questionnaires: Patients will complete surveys before the treatment period, immediately after the treatment period, and four weeks post-treatment.

MRI & EEG: Patients will undergo brain imaging (MRI) and brain wave (EEG) recordings before and after the treatment period.

Adverse Effects Diary: Patients will maintain a daily log of any side effects experienced during the treatment period.

The study aims to assess the feasibility, safety, and effectiveness of this combined treatment approach and to examine its effects on underlying brain processes related to clinical outcomes.

DETAILED DESCRIPTION:
This study aims to explore the combination of specialized inpatient care for Obsessive-Compulsive Disorder (OCD) with treatment using repetitive Transcranial Magnetic Stimulation (rTMS) in patients diagnosed with OCD. Specifically, the investigators seek to assess the feasibility, desirability, and tolerability of this combined approach, as well as its clinical and neural effects.

The study protocol consists of three arms. All arms include Exposure and Response Prevention (ERP), an established psychotherapeutic treatment for OCD. Two arms will investigate two different types of rTMS: conventional deep TMS (dTMS) and intermittent theta burst stimulation (iTBS). Both rTMS treatments will be administered using an accelerated protocol, involving four sessions per day. The third arm consists of ERP without any form of neuromodulation (i.e., treatment-as-usual).

Study Design:

This is a randomized clinical trial (RCT) evaluating the feasibility, efficacy, safety, and suitability of the two types of accelerated rTMS protocols, in addition to ERP therapy in patients with OCD. The study also aims to investigate the neural mechanisms underlying these treatment approaches.

Patients will be randomly assigned by a computer program to one of three treatment groups. All groups will receive ERP. Two groups will receive either iTBS or dTMS combined with ERP, and the third group will receive ERP without rTMS.

Participant Requirements:

Questionnaires: Completion of surveys before treatment, immediately after treatment, and four weeks post-treatment.

MRI & EEG: Undergo functional and structural brain imaging (MRI) and high-definition electroencephalography (hdEEG) before and after the treatment period.

Adverse Effects Diary: Maintain a daily log of any side effects experienced during the treatment period.

Study Duration:

The total expected duration of participation is ten weeks. Magnetic stimulation treatment will take place over two weeks, within a standard hospitalization of twelve weeks in an OCD inpatient department. Participation does not require additional hospital visits compared to usual treatment.

Study Location:

The study will be conducted at UZ Gent, Building K12F, Corneel Heymanslaan 10, 9000 Ghent, Belgium. A total of 60 patients will participate, with 40 patients receiving rTMS treatment. All procedures will take place within Belgium.

Participant Involvement:

During the twelve-week hospitalization, rTMS treatment will commence approximately two weeks after admission. The initial two-week period allows for familiarization with the department and ERP therapy. Prior to inclusion, eligibility will be assessed through a 60-minute consultation, a semi-structured diagnostic interview (MINI-5), and a structured assessment of OCD symptoms (Y-BOCS symptom checklist) to identify any exclusion criteria or contraindications.

Eligible patients will undergo two brain imaging procedures: functional and structural MRI and hdEEG. Additionally, five questionnaires will be administered collectively.

The rTMS protocol will then be implemented over a two-week period, with four sessions per day, four days per week, totaling 32 sessions. During this period, patients will complete a daily adverse effects questionnaire. Immediately after treatment, post-treatment assessments will include questionnaires and repeated fMRI and hdEEG scans. Four weeks later, follow-up questionnaires assessing OCD symptoms and related measures will be completed.

Certain visits and procedures described in the study will be part of standard care at the hospital, while others are specific to the research protocol. Throughout the twelve-week hospitalization, all groups will receive standard care, including medication optimization and evidence-based psychotherapeutic interventions for OCD. rTMS will be offered as an adjunctive treatment to this standard care.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65
* Hospitalization for Obsessive-Compulsive Disorder (OCD)
* Participation in Exposure and Response Prevention Therapy
* Significant OCD, as measured by a Y-BOCS score of 20 or higher (moderate to severe OCD symptoms)

Exclusion Criteria:

* Acute suicidality: Individuals presenting with current suicidal ideation or behavior are excluded to ensure participant safety.
* Psychotic disorder: patients with active psychotic disorders are excluded due to the complexity of their condition and potential interactions with the study protocol.
* Current substance use disorder: active substance use disorders are exclusionary to prevent confounding effects on study outcomes.
* Deep Brain Stimulation (DBS) for OCD: participants with an implanted DBS device for OCD are excluded due to potential interference with the study's interventions and safety concerns.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-25 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-Reported Severity of Adverse Effects [Safety] | From start to end of rTMS treatment period (2 weeks)
  Severity of specific adverse effects (e.g., headache, tooth pain, scalp discomfort, fatigue, etc.) will be assessed daily using a visual analogue scale (VAS) ranging from 0 (not at all) to 10 (extremely severe). Scores will be collected daily for the duration of the treatment.
  Unit of Measure: VAS score (0-10) per adverse effect
Incidence of Any Self-Reported Adverse Effect [Safety] | From start to end of rTMS treatment period (2 weeks)
  Occurrence of any self-reported adverse effect (i.e., VAS > 0 for any symptom) during the rTMS treatment period.
  Unit of Measure: Number of participants reporting ≥1 adverse effect
Participant Retention Rate [Feasibility] | From enrollment to end of treatment (approximately 2 weeks of rTMS)
  Percentage of participants who complete the full rTMS treatment protocol (32 sessions over 2 weeks) out of those who consented and were randomized.
  Unit of Measure: Percentage of participants completing protocol

SECONDARY OUTCOMES:
Functional MRI-Based Resting-State Functional Connectivity | Before and after each treatment arm (2 weeks).
  Resting-state functional MRI (rs-fMRI) will be used to assess changes in intrinsic brain network connectivity. Whole-brain and region-of-interest (ROI) connectivity analyses will be performed.
  Unit of Measure: Change in functional connectivity (Fisher z-scores or correlation coefficients) between selected brain regions
Structural MRI-Based Grey Matter Volume | Before and after each treatment arm (2 weeks).
  Structural MRI scans will be used to estimate grey matter volume in regions implicated in OCD and rTMS target. Voxel-based morphometry and region-specific volumetric analyses will be performed.
  Unit of Measure: Change in grey matter volume in specified regions
DTI-Based White Matter Microstructure | Before and after each treatment arm (2 weeks).
  Diffusion Tensor Imaging (DTI) will be used to assess white matter integrity through metrics such as fractional anisotropy (FA) and mean diffusivity (MD). Analyses will focus on tracts implicated in OCD and rTMS targets.
  Unit of Measure: Change in DTI metric values in specified white matter tracts.
ASL-Based Resting Cerebral Blood Flow | Before and after each treatment arm (2 weeks).
  Arterial Spin Labeling (ASL) MRI will be used to quantify resting-state cerebral blood flow (CBF) in regions relevant to OCD pathophysiology and rTMS target. Region-of-interest and whole-brain voxelwise analyses will be performed.
  Unit of Measure: Change in CBF in specified brain regions.
EEG-Based Resting-State Oscillatory Power | Before and after each treatment arm (2 weeks).
  High-definition EEG will be used to quantify resting-state oscillatory activity in standard frequency bands (delta, theta, alpha, beta, gamma). Unit of Measure: Change in spectral power per frequency band and region.
EEG-Based Resting-State Functional Connectivity | Before and after each treatment arm (2 weeks).
  Functional connectivity will be assessed using phase- and coherence-based metrics to evaluate connectivity between cortical regions of interest. Unit of Measure: Change in connectivity strength.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Baeken, PhD. MD. Psychiatry, Principal Investigator — UZ GENT
Locations (1):
- UZ Gent, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- See also: Related Info — http://gheplab.ugent.be